CLINICAL TRIAL: NCT07322731
Title: The Effect of Massage on Sleep Quality, Stress, Comfort, and Vital Signs in Preterm Infants: A Randomized Controlled Trial
Brief Title: The Effect of Massage on Sleep Quality, Stress, Comfort, and Vital Signs in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Rıdvan Akdogan, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUZUNCU_YIL_UNIVERSITY_NICU
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Premature Infants; Sleep Quality; İnfant Stress; İnfant Comfort; Vital Signs; NICU
Keywords: Preterm infants; neonatal massage; NICU; sleep quality; stress reduction; comfort; vital signs
MeSH Terms: conditions — Premature Birth; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the intervention group, which receives massage therapy, or the control group, which receives standard care. Randomization is performed using the Urn method. Each participant is assigned to only one group (parallel design). The intervention is applied three times daily for 15 minutes over three consecutive days.
Masking Description: No masking; open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Preterm infants receiving massage therapy three times daily for 15 minutes over 3 days, in addition to standard care.
  Interventions: Other: Infant Massage Therapy
- Control - Standard Care (No Intervention): Preterm infants receiving standard care only, without massage intervention.

INTERVENTIONS:
Other: Infant Massage Therapy — Preterm infants receive a standardized massage therapy protocol three times daily for 15 minutes over 3 days. The massage is applied by a trained nurse and includes legs, arms, and back following a structured sequence.
  Arms: Experimental Group

SUMMARY:
This randomized controlled trial investigates the effects of massage therapy on sleep quality, stress, comfort, and vital signs in preterm infants (gestational age 35-37 weeks) admitted to the Neonatal Intensive Care Unit (NICU) at Van YYU Training and Research Hospital. Infants in the intervention group will receive a 15-minute massage three times a day for three consecutive days, while the control group will receive standard care. Data will be collected using the Premature Infant Comfort Scale, Neonatal Stress Scale, actigraphy for sleep monitoring, and vital sign measurements. The study aims to determine whether massage therapy can improve the overall well-being and development of preterm infants in NICU settings.

DETAILED DESCRIPTION:
This randomized controlled study evaluates the impact of massage therapy on preterm infants' sleep quality, stress levels, comfort, and vital signs in the Neonatal Intensive Care Unit (NICU) at Van YYU Training and Research Hospital. Infants born between 35 and 37 weeks of gestation and meeting inclusion criteria will be randomly assigned to either an intervention group receiving massage or a control group receiving standard care.

The intervention consists of a 15-minute massage administered three times daily for three consecutive days by a trained researcher. Massage includes gentle stroking and circular movements of the legs, arms, back, and hands, following a standardized protocol. Physiological parameters (heart rate, respiratory rate, blood pressure, oxygen saturation), sleep patterns (using actigraphy and chronometer), and behavioral assessments using the Premature Infant Comfort Scale and Neonatal Stress Scale will be recorded before and after the intervention.

Data will be analyzed using SPSS version 25. Group homogeneity will be assessed with chi-square or Fisher's exact tests, within-group comparisons with paired t-tests, and between-group comparisons with independent t-tests. Significance will be set at p < 0.05. This study aims to provide evidence on the efficacy of massage therapy as a non-pharmacological intervention to improve preterm infants' comfort, reduce stress, and enhance sleep quality in NICU settings.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 35-37 weeks gestational age.
* Admitted to the neonatal intensive care unit (NICU).
* Medically stable and cleared for massage therapy by neonatologist.
* Parental/guardian consent obtained.

Exclusion Criteria:

* Infants with congenital anomalies or major medical complications.
* Infants requiring mechanical ventilation or intensive respiratory support.
* Infants with known neurological disorders.
* Parental/guardian refusal or inability to participate.

Ages: 35 Months to 37 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality of Preterm Infants | Measured daily over 3 days of massage intervention
  Sleep duration and awakenings assessed using actigraphy and researcher observation before and after massage sessions.

SECONDARY OUTCOMES:
Infant Comfort Level | Assessed before first massage and after last massage session (Day 3)
  Measured using Premature Infant Comfort Scale , higher scores indicate lower comfort.
Infant Stress Levels | Assessed before first massage and after last massage session (Day 3)
  Measured using Neonatal Stress Scale; higher scores indicate greater stress.
Heart Rate of Preterm Infants During Massage Therapy | Baseline (prior to the first massage session) and immediately after each massage session over 3 days
  Heart rate will be measured using a bedside monitor as an indicator of physiological response to massage therapy. Unit of measure: beats per minute (bpm).
Respiratory Rate of Preterm Infants During Massage Therapy | Baseline (prior to the first massage session) and immediately after each massage session over 3 days
  Respiratory rate will be measured using a bedside monitor as an indicator of physiological response to massage therapy. The outcome will be expressed as breaths per minute.
Oxygen Saturation of Preterm Infants During Massage Therapy | Baseline (prior to the first massage session) and immediately after each massage session over 3 days
  Oxygen saturation will be measured noninvasively using pulse oximetry to assess physiological response to massage therapy. The outcome will be expressed as percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Van Regional Training and Research Hospital, Van, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data, along with the study protocol and statistical analysis plan, will be made available upon reasonable request to researchers. Data will be accessible starting 6 months after publication of the primary results and will remain available for 5 years.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting documents will be available beginning six months after the publication of the primary study results and will remain accessible for a period of five years.
Access Criteria: Qualified researchers may request access to de-identified individual participant data, the study protocol, and statistical analysis plan. Requests must be submitted via email to the corresponding author, and data will be shared under a data use agreement.